CLINICAL TRIAL: NCT03765723
Title: Prediction Model of Acute Postoperative Pain in Bilateral Total Knee Replacement Arthroplasty Patient: Multivariable Model Including "Surgical History Within 2 Weeks" as a Predictive Factor
Brief Title: Prediction Model of Acute Postoperative Pain in Bilateral Total Knee Replacement Arthroplasty Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: SNUMR2-1
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Arthritis Knee; Anesthesia; Arthropathy of Knee
Keywords: TKRA; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to predict risk factors of acute postoperative pain of the patients undergoing Total Knee Replacement Arthroplasty(TKRA).

DETAILED DESCRIPTION:
Patients undergoing bilateral TKRA are recruited. The time interval between the surgery of each leg is within 2 weeks. Before each surgery, patients will be asked to conduct questionnaires of Hospital Anxiety and Depression Scale(HADS) and Pain Catastrophizing Scale(PCS). In addition, the patients will have their preoperative knee pain(measured by Knee injury and Osteoarthritis Outcome Score), preoperative pain in other sites, expectation of postoperative pain(measured by Numerical Rating Scale), and morbidity of diabetic neuropathy recorded. Demographic factors including age, sex, and BMI of patients will be collected. Twenty four and forty eight hours after completion of the surgery, each patient will be asked to report thier acute postoperative pain on Numerical Rating Scale.

This study aims to find out risk factors of acute postoperative pain, including identical surgical history within 2 weeks, in patients undergoing bilateral TKRA.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients undergoing bilateral TKRA with spinal anesthesia
* 2) patients who have their second TKRA in one leg within 2 weeks after their first TKRA in the other leg.
* 3) patients who are classified to the state of ASA physical status classification system Ⅰ,Ⅱ, or Ⅲ.

Exclusion Criteria:

* 1) patients incapable of communication

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing bilateral TKRA will be recruited from the patients in Seoul National University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute post operative pain | 24 hours
  Acute post operative pain is recorded on Numerical Rating Scale(a pain scale ranging from 0 to 10. the higher number means the higher pain) at rest in an attempt to bent knee.
Acute post operative pain | 48 hours
  Acute post operative pain is recorded on NRS(a pain scale ranging from 0 to 10. the higher number means the higher pain) at rest in an attempt to bent knee.
Consumption of analgesics | 48 hours
  Cumulative consumption of Patient-Controlled Analgesia(PCA) and rescue analgesics is recorded.

SECONDARY OUTCOMES:
Preoperative anxiety and depression | one day before the surgery: 20 hours before the surgery
  Before undergoing TKRA of each leg, patients' preoperative anxiety and depression is recorded on Hospital Anxiety and Depression Scale(HADS) total score.
  HADS is an instrument for screening for clinically significant anxiety and depression in patients attending a general medical clinic. The scale consists of two subscales: anxiety subscale and depression subscale. Each subscale has seven items and each items are answered by the patient on a four point(0-3) response categories so the possible score ranges from 0 to 21 for anxiety and 0 to 21 for depression(summation). A score of 0 to 7 for either subscale could be regarded as being in normal range, a score of 8-10 being suggestive of the presence of the mood disorder, and a score of 11 or higher indicating probable presence of the respective state.
Pain catastrophizing level | one day before the surgery: 20 hours before the surgery
  Before undergoing TKRA of each leg, patients' pain catastrophizing level is recorded on Pain Catastrophizing Scale(PCS) total score.
  PCS is a thirteen-item instrument to assess patient's catastrophizing on pain experience. The scale consists of three subscales: rumination(4 items), magnification(3 items), and helplessness(4 items). For each items, patients are asked to response on a five point(0-4) categories so the total score is ranging from 0 to 52(summation). A total PCS score of 30 is considered cut-off scores for clinically relevant levels of catastrophizing. The higher score represents high level of catastrophizing.
Preoperative knee pain | one day before the surgery: 20 hours before the surgery
  Before undergoing TKRA of each leg, patients' preoperative knee pain is recorded on Knee injury and Osteoarthritis Outcome Score(KOOS) pain subscale score.
  KOOS is an instrument to assess pain, symptoms, activities of daily living, sport and recreation function, and knee related quality of life of the patients with ligament injury, meniscus injury, or post traumatic osteoarthritis. A pain subscale of KOOS consists of nine items to assess the level of pain in knee, each item being scored from 0 to 4. A total score of pain subscale ranges from 0 to 36(summation). In this raw scale score on pain, the higher score means the higher level of pain.
Preoperative pain in other sites | one day before the surgery: 20 hours before the surgery
  Before undergoing TKRA of each leg, patient's preoperative pain in other sites is recorded on NRS(a pain scale ranging from 0 to 10. the higher number means the higher pain).
Pain expectation of acute postoperative pain | one day before the surgery: 20 hours before the surgery
  Before undergoing TKRA of each leg, patient's pain expectation of acute postoperative pain is recorded on NRS(a pain scale ranging from 0 to 10. the higher number means the higher pain).
Diabetic neuropathy | one day before the surgery: 20 hours before the surgery
  Patient's diabetic neuropathy is recorded by searching electronic medical records or directly asked.
Demographic data | one day before the surgery: 20 hours before the surgery
  Patient's age, sex, and BMI is recorded by searching electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: JINTAE KIM, M.D. / Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No